CLINICAL TRIAL: NCT00389259
Title: Scopolamine Treatment for Patients With Organophosphate Poisoning - a Randomized, Double Blind, Placebo-Controlled Study.
Brief Title: Scopolamine Treatment for Patients With Organophosphate Poisoning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Israeli MOH (Unknown); International Diabetes Federation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70/04*1
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2010-03

CONDITIONS: Neurotoxicity Syndromes
Keywords: Insecticides; Organophosphate; Scopolamine; randomized control study; Organophosphate or carbamate intoxication
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): IV Scopolamine 0.25mg in adults and 0.006mg/kg in children Q4h
  Interventions: Drug: Placebo
- B (Placebo Comparator): IV Look alike drug Q 4h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — IV placebo q4h

SUMMARY:
Organophosphate (OP) compounds are a major threat as chemical warfare agents or in terrorist act. OPs are also the active ingredient of many insecticides. Ingestion of insecticides is a common cause of death among people who commit suicide in developing countries. OPs poisoning also frequently occurs after accidental exposure to agricultural OPs and in children as a result of unintentional ingestion.

The use of competitive inhibitors of acetylcholine other than atropine for patient with organophosphate (OP) poisoning is controversial. Because scopolamines' ability to cross the blood brain barrier is better than atropine, it has been suggested that scopolamine should be used OP poisoned patients who have central nervous system (CNS) manifestations. However there is controversy regarding its potential benefit in the treatment of organophosphate poisoning in humans. To the best of our knowledge there are no randomised controlled studies on the use of scopolamine in humans. This prospective randomised controlled study is aimed to determine whether adding scopolamine to the standard treatment of atropine and oximes in patients with CNS symptoms of OP poisoning improve the outcome.

DETAILED DESCRIPTION:
Objective: to determine whether adding scopolamine to the standard treatment of atropine and oximes improve the outcome of patients with OP poisoning and CNS manifestations. Design: A multi-center, randomized, double blind, placebo controlled study. Setting: Emergency Departments & Intensive Care Units in Israel. Participants: Patients 2 -60 years old with acute OP poisoning and CNS manifestations. Interventions: In addition to standard treatment with atropine and obidoxime, eligible patients will be randomly assigned to one of two treatment groups, scopolamine group, and placebo group (both given in the same volume). Scopolamine will be given IM or IV in a dose of 0.25mg for adults and 0.006mg/kg for children every 4 hours. At least three doses of scopolamine (or placebo) will be given. The medical staff will be blinded to the treatment given. Main outcome measures: Improvement in neurological status, duration of seizures and number of days on ventilator. Data analysis: The main outcome measures, will be compared using the Student's t-test or the Mann-Whitney tests as appropriate. The *2 or Fisher Exact tests, as appropriate, will be used for comparisons of categorical variables. We will use multiple logistic regression to examine the extent to which variables predict success or failure of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2- 60 years
* At least two of the following three criteria:

  * Known exposure to an organophosphate or carbamate insecticide in the last 72 hours.
  * Symptoms and signs typical to organophosphate poisoning involving at least two systems (gastrointestinal, respiratory, skin, eyes,) See appendix
  * Low levels of plasma butyrylcholinesterase (less than 50% of the lower normal range )
* CNS involvement in the first 72 hours after exposure: determined by finding at least one of the following major criteria or at least two of the minor criteria

Major criteria for CNS involvement:

* Seizures
* Extrapyramidal or Parkinson like symptoms
* Decreased level of consciousness (GCS< 12)

Minor criteria for CNS involvement:

* GCS 14-12
* Confusion
* Hallucinations

Exclusion Criteria:

* Hypersensitivity to scopolamine
* Glaucoma, narrow-angle (angle-closure)
* Tachyarrhythmias, congestive heart failure
* Obstructive gastrointestinal disease
* Myasthenia Gravis
* Reflux esophagitis
* Ulcerative colitis
* Known obstructive uropathy
* Pregnancy
* Patient or legal guardian unable to give informed consent (see comment under ethics)
* Severe co-morbidity (multi-trauma, advanced cancer, etc)

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in neurological status as measured by the Glasgow Coma Scale | 1 week
Duration of seizures. | 1 week
Number of days on ventilator | 1 week

SECONDARY OUTCOMES:
Total cumulative dose of atropine | 1 week
Need for benzodiazepines | 1 week
Number of days in the ICU | 2 weeks
Adverse effects and complications | 2 weeks
Neurological assessment at discharge | 2 weeks
Neurological assessment 3 month after the exposure | 3 month
Neuro-cognitive assessment at 3 month | 3 month
Survival at 24 hours | 24 hours
Survival to discharge | 4 weeks
Number of days in hospital | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eran Kozer, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Rambam Hospital, Haifa, Israel